CLINICAL TRIAL: NCT05040009
Title: Foot Care and Footwear Assessment in Diabetic Patients and Its Relation to Diabetic Complications.
Brief Title: Foot Care Assessment and Relation to Diabetic Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Paula Rofaeel Sedky, Assistant lecturer Faculty of Medicine, ِِAssiut University, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Foot care assessment in DM
Record Dates: First submitted 2021-08-22; First posted 2021-09-10 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate and high risk patient with integrated foot care program (Active Comparator): Integrated foot care program will be applied to moderate and high-risk patients for diabetic foot with follow up after 6-12 months
  1. Regular foot care and examination by an adequately trained professional: -
  2. Structured education
  3. Adequate footwear
  4. Foot-related exercises and weight-bearing activity.
  5. Foot examination and screening every 4 months in moderate risk and 2 months in high-risk patient for diabetic foot.
  6. Instructions about foot self-management
  Interventions: Behavioral: integrated foot care program
- moderate and high risk patient with conventional treatment (No Intervention): conventional treatment will be applied to moderate and high-risk patients for diabetic foot with follow up after 6-12 months.

INTERVENTIONS:
Behavioral: integrated foot care program — 1. Regular foot care and examination by an adequately trained professional: -
  2. Structured education:
  Educational modality will be provided to patients in a structured way. This will take many forms: one-to-one verbal education session last around 30 min motivational interviewing, video education, booklets, pictorial education via animated drawing or descriptive images structured foot care education consists of information on:
  1. Foot ulcers and their consequences
  2. Preventative foot self-care behaviors
  3. Wearing adequately protective footwear
  4. Undergoing regular foot checks
  5. Practicing proper foot hygiene
  6. Seeking professional help in a timely manner after identifying a foot problem
  3-Adequate footwear 4-Foot-related exercises and weight-bearing activity 5-Foot examination and screening 6- Instructions about foot self-management
  Arms: moderate and high risk patient with integrated foot care program

SUMMARY:
Screening for diabetic foot in patients attending at Diabetic center at Assiut university and its relations to diabetic microvascular complications (nephropathy, neuropathy and retinopathy) and macrovascular complications (stroke , myocardial infarction and peripheral arterial diseases).

Footwear assessment in diabetic patient. Evaluation of integrated foot care program in moderate and high-risk patients for diabetic foot.

Evaluation of knowledge and practice of diabetic foot

DETAILED DESCRIPTION:
The International Diabetes Federation (IDF) has identified Egypt as the ninth leading country in the world for the number of patients with T2D. The prevalence of T2D in Egypt was almost tripled over the last 2 decades. This sharp rise could be attributed to either an increased pattern of the traditional risk factors for T2D such as obesity and physical inactivity and change in eating pattern or other risk factors unique to Egypt .

Diabetic foot complications are the most common cause of non-traumatic lower extremity amputations in the industrialized world, may cause death or physical and psychical disability, has a great impact on quality of life, and represents a high cost for society ( .

The term diabetic foot encompasses any lesion in the feet: infection, ulcer, and destruction of deep tissues occurring as the result of diabetes and its complications .

The absence of symptoms in a person with diabetes does not exclude foot disease; they may have asymptomatic neuropathy, peripheral artery disease, pre-ulcerative signs, or even an ulcer.

Every diabetic patient will be subjected to

1. Medical history.
2. Therapeutic history: Antidiabetic drugs (type, duration), other medications for obesity, hypertension and dyslipidemia
3. Complete physical examination.
4. The following work up;

   * Knowledge questionnaire developed by Hasnain and colleagues and the Nottingham Assessment of Functional Foot Care (NAFFC) .
   * Screening for diabetic foot .
   * Fundus examination
   * ECG
   * The following investigations: Alb/cre ration, HBA1c, lipid profile, blood urea, serum creatinine
   * Abdominal ultrasound
   * Ankle brachial index (ABI)
5. Integrated foot care program will be applied to moderate and high-risk patients for diabetic foot with follow up after 6-12 months vs conventional education

ELIGIBILITY:
Inclusion Criteria:

Adult patient with diabetic mellitus

Exclusion Criteria:

Major amputation of lower limbs. End stage organ failure. Diabetic patient less than 18 years or more than 75. Pregnant diabetic women. Connective tissue disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Integrated foot care program in moderate and high-risk patients for diabetic foot versus conventional treatment | 6 to 12 month
  moderate and high risk patients for diabetic foot will undergo integrated program vs conventional treatment as regard ulcer healing and recurrence
Evaluation of knowledge and practice of diabetic foot using questionnaire developed by Hasnain and colleagues and the Nottingham Assessment of Functional Foot Care (NAFFC) | baseline
  knowledge and practice are assessed using questionnaire developed by Hasnain and colleagues and the Nottingham Assessment of Functional Foot Care (NAFFC)
Screening for diabetic foot and diabetic complication in patients attending at Diabetic center | baseline
  Screening for diabetic foot in patients attending at Diabetic centre at Assiut university according to IWGDF guidelines Every diabetic patient will be subjected to Fundus examination ECG The following investigations: Alb/creatinine ratio, HBA1c, lipid profile, blood urea, serum creatinine Abdominal ultrasound Ankle brachial index (ABI)

CONTACTS AND LOCATIONS:
Locations (1):
- Paula Rofaeel, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Hegazi R, El-Gamal M, Abdel-Hady N, Hamdy O. Epidemiology of and Risk Factors for Type 2 Diabetes in Egypt. Ann Glob Health. 2015 Nov-Dec;81(6):814-20. doi: 10.1016/j.aogh.2015.12.011. PMID 27108148
- [Background] Prompers L, Schaper N, Apelqvist J, Edmonds M, Jude E, Mauricio D, Uccioli L, Urbancic V, Bakker K, Holstein P, Jirkovska A, Piaggesi A, Ragnarson-Tennvall G, Reike H, Spraul M, Van Acker K, Van Baal J, Van Merode F, Ferreira I, Huijberts M. Prediction of outcome in individuals with diabetic foot ulcers: focus on the differences between individuals with and without peripheral arterial disease. The EURODIALE Study. Diabetologia. 2008 May;51(5):747-55. doi: 10.1007/s00125-008-0940-0. Epub 2008 Feb 23. PMID 18297261
- [Background] Apelqvist J, Bakker K, van Houtum WH, Nabuurs-Franssen MH, Schaper NC. International consensus and practical guidelines on the management and the prevention of the diabetic foot. International Working Group on the Diabetic Foot. Diabetes Metab Res Rev. 2000 Sep-Oct;16 Suppl 1:S84-92. doi: 10.1002/1520-7560(200009/10)16:1+3.0.co;2-s. PMID 11054895
- [Background] Hasnain S, Sheikh NH. Knowledge and practices regarding foot care in diabetic patients visiting diabetic clinic in Jinnah Hospital, Lahore. J Pak Med Assoc. 2009 Oct;59(10):687-90. PMID 19813683